CLINICAL TRIAL: NCT05559385
Title: Is Robot-Assisted System Effective for the Maximization of Upper Extremity Motor Recovery in Intensive Body Rehabilitation Following a Stroke
Brief Title: Is Robot-Assisted Therapy Effective for the Upper Extremity Following a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emresenocak (Other)
Responsible Party: Sponsor-Investigator, Emresenocak, Research Assisstant, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2021.168
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Stroke
Keywords: Robotic Rehabilitation; Conventional Rehabilitation; Intensıve Trunk Rehabilitation; Motor Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled (One group received Robotic Rehabilitation, other group received conventional rehabilitation)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Rehabilitation Group (Experimental): The standardized ITR program was applied to both groups for 60 minutes a day, five days a week, for six weeks. The ITR program included exercises of abdominal strengthening, controlled pelvic movements, bridging, trunk lateral flexion and rotation, reaching forward, and push-ups with a Swiss Ball. This group received a robotic rehabilitation program for the upper extremity with a Houston Bionics ExoRehab X brand/model device. This device has no motor force of repulsion or attraction. Patients initiate and maintain their movements during the exercise. The device supports the patient's active movement and allows extensive movement repetition.
  Before starting robotic rehabilitation, the patient was seated upright on the platform. The games were projected onto a 43-inch television screen. The exercise program was planned to include upper extremity movements in all directions.
  Interventions: Device: Robot-Assissted Therapy
- Conventional Rehabilitation Group (Active Comparator): The standardized ITR program was applied to both groups for 60 minutes a day, five days a week, for six weeks. During this period, lower extremity rehabilitation was added if needed in addition to trunk rehabilitation. Exercises for the lower extremities were applied according to the patient's individual needs. The ITR program included exercises of abdominal strengthening, controlled pelvic movements, bridging, trunk lateral flexion and rotation, reaching forward and sideways, and push-ups with a Swiss Ball.
  CR applied after the ITR program consisted of an individualized rehabilitation program for the upper extremities. These rehabilitation programs generally included activities for functional purposes (dressing, object manipulation, reaching, cup holding, range of motion, strengthening, weight-bearing, etc.). The treatment program was applied five days a week for six weeks, with the session duration limited to 60 minutes.
  Interventions: Procedure: Conventional Rehabilitation

INTERVENTIONS:
Device: Robot-Assissted Therapy — Houston Bionics ExoRehab X brand/model device was used for improving the upper extremity in subacute stroke.
  Arms: Robotic Rehabilitation Group
Procedure: Conventional Rehabilitation — It is an upper extremity rehabilitation program prepared in line with individual needs.
  Arms: Conventional Rehabilitation Group

SUMMARY:
The aim of this study was to investigate the effects on upper-limb motor function of the addition of robotic rehabilitation (RR) and conventional rehabilitation (CR) treatments to intensive trunk rehabilitation (ITR).

A total of 41 subacute stroke patients were randomly allocated to two groups: RR and CR. Both groups received the same ITR procedure (6x5x60 weeks/days/minutes). Following ITR, a robot-assisted rehabilitation program of 60 minutes, five days a week, for six weeks, was applied to the RR group, and an individualized upper extremity rehabilitation program to the CR group. Evaluations were made at baseline and after six weeks using the Trunk Impairment Scale (TIS), Fugl-Meyer Upper Extremity Motor Evaluation Scale (FMA-UE), and Wolf Motor Function Test (WMFT).

DETAILED DESCRIPTION:
Assessments:

- Demographic Data Form: The researchers created a form to include the information on age, gender, stroke onset date, lesion type, affected side, and dominant extremity.

- Fugl-Meyer Upper Extremity Assessment: This disease-specific scale was created as an objective motor impairment scale to assess recovery in post-stroke hemiplegic patients (18). It includes subsections that assess joint movements, coordination, and reflex activities related to the shoulder, elbow, forearm, wrist, and hand. The maximum score that can be obtained is 66, with a high score indicating good motor condition. The affected upper extremities are assessed with the subject in a seated position.

- Wolf Motor Function Test: This test was created to evaluate the motor ability of the upper extremity (19). The test consists of 17 items, 15 of which are related to the fields of functional skill and performance time, and 2 to muscle strength (20). The total score is used for the functional ability of the patients. The two items of muscle strength evaluation were not used in this study.

- Trunk Impairment Scale: This scale evaluates static and dynamic sitting balance and trunk coordination with seventeen items. The total score ranges from 0 - 23 points, with a higher score indicating better performance. The test-retest and inter-rater reliability coefficients of the scale have been shown to be 0.85-0.99 (21).

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85 years and having had a stroke in the last six months,
* Mini-Mental State Assessment score >20,
* Able to sit safely,
* No neglect issue,
* Fugl-Meyer Upper Extremity Assessment score <58.

Exclusion Criteria:

* Modified Ashworth Scale >2,
* Severe reduction in visual acuity,
* Participation in another rehabilitation program,
* Subluxation or pain in the shoulder region.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Assessment: | At the baseline
  This disease-specific scale was created as an objective motor impairment scale to assess recovery in post-stroke hemiplegic patients. It includes subsections that assess joint movements, coordination, and reflex activities related to the shoulder, elbow, forearm, wrist, and hand. The maximum score that can be obtained is 66, with a high score indicating good motor condition.
Fugl-Meyer Upper Extremity Assessment: | At the end of the 6th week
  This disease-specific scale was created as an objective motor impairment scale to assess recovery in post-stroke hemiplegic patients. It includes subsections that assess joint movements, coordination, and reflex activities related to the shoulder, elbow, forearm, wrist, and hand. The maximum score that can be obtained is 66, with a high score indicating good motor condition.

SECONDARY OUTCOMES:
Demographic Data Form | At the baseline
  Demographic Characteristics
- Wolf Motor Function Test: | At the baseline
  This test was created to evaluate the motor ability of the upper extremity. The test consists of 17 items, 15 of which are related to the fields of functional skill and performance time, and 2 to muscle strength (20). The two items of muscle strength evaluation were not used in this study. A high score indicates fine motor ability.
- Wolf Motor Function Test: | At the end of the 6th week
  This test was created to evaluate the motor ability of the upper extremity. The test consists of 17 items, 15 of which are related to the fields of functional skill and performance time, and 2 to muscle strength (20). The two items of muscle strength evaluation were not used in this study. A high score indicates fine motor ability.
Trunk Impairment Scale | At the baseline
  This scale evaluates static and dynamic sitting balance, and trunk coordination with seventeen items. The total score ranges from 0 - 23 points, with a higher score indicating better performance.
Trunk Impairment Scale | At the end of the 6th week
  This scale evaluates static and dynamic sitting balance, and trunk coordination with seventeen items. The total score ranges from 0 - 23 points, with a higher score indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yildiz Ozer, PhD, Study Director — Marmara University; Adem Aktürk, PhD, Principal Investigator — Gelişim University; Elif Korkut, PhD, Principal Investigator — Bağcılar Education and Research Hospital
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Senocak E, Korkut E, Akturk A, Ozer AY. Is the robotic rehabilitation that is added to intensive body rehabilitation effective for maximization of upper extremity motor recovery following a stroke? A randomized controlled study. Neurol Sci. 2023 Aug;44(8):2835-2843. doi: 10.1007/s10072-023-06739-3. Epub 2023 Mar 10. PMID 36897464